CLINICAL TRIAL: NCT00543647
Title: A Double-blind, Cross-over, Placebo-controlled Study Evaluating the Effect of Fenofibrate 160 mg Tablets on Glomerular Filtration Rate and Other Renal Function Test in Healthy Subjects
Brief Title: Effect of Fenofibrate on Kidney Function: a Six-week Randomized Cross-over Trial in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CFEN 0201
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2007-10

CONDITIONS: Healthy Volunteers
Keywords: Fenofibrate; Glomerular filtration rate; inulin clearance; creatinine; healthy volunteers; cross-over
MeSH Terms: interventions — Fenofibrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate 160 mg tablet
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate 160 mg tablet
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study was to test the effect of fenofibrate treatment on glomerular filtration rate (GFR), kidney hemodynamics and tubular function in middle-aged subjects with normal kidney function to further investigate the increase in creatinine levels observed in fenofibrate-treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age: 30-60 years old
* Subjects with normal renal function as documented by: Plasma creatinine < 130 µmol/L, AND Cockcroft & Gault creatinine clearance (Co Cr CL) >80 ml/min
* Certified as normal by a comprehensive medical assessment and laboratory investigations the results of which are within the normal range /or clinically acceptable for the present subjects and who have a negative urinary screen for drugs of abuse.
* Written informed consent

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m² or <18 kg/m².
* Pregnant, breast-feeding, or woman with child bearing potential without a reliable method of contraception.
* Having received an investigational drug in the last 90 days before date of inclusion.
* With known hypersensitivity to fibrates.
* Unable or unwilling to comply with the protocol, or likely to leave the study before its completion.
* Who would undertake important change in physical exercise or vigorous sport competitions during the study period.
* Drug therapies are not permitted during the study, except contraceptive pill when applicable, with the exception of occasional use of paracetamol.
* Any administration of treatment, which could bring about induction or inhibition of hepatic microsomal enzymes within 3 months of the study start.
* Diabetes mellitus, Heart diseases, Kidney diseases, hypertension, asthma, Liver diseases, Chronic pancreatitis, or identified risk or known history of acute pancreatitis, Known cholelithiasis without cholecystectomy, ASAT and/or ALAT > 1.3 times ULN, Gastric or peptic ulcer or intestinal diseases, Musculoskeletal diseases or increased CK > 1.0 times ULN, History of neoplasm, Mental illness, Regular user of sedatives, hypnotics, tranquillisers or any other addictive agents or who are known to be prone to alcohol abuse (i.e. history or evidence of acute abuse), or alcohol intake >14 units per week (unit = ½ pint of beer, 1 glass of wine, 2,5 cl standard spirits), or heavy smokers (>10 cigarettes/day), or excessive drinker of tea, coffee and/or beverages containing caffeine (>8 cups/day), Blood donor with recent donation (in the three months preceding the initiation of the study) or would make blood donations during the study, Blood transfusion or administration of blood-derived products, in the year preceding the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-08; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) assessed by the measure of inulin clearance | After two periods of 6 weeks treatment (fenofibrate and placebo in cross-over) separated by a 6wks wash out

SECONDARY OUTCOMES:
GFR evaluated by raw values of plasma creatinine and cystatin C levels | before and after each treatment period
Renal haemodynamics evaluated by raw values of renal plasma and blood flows | before and after each treatment period
Tubular function: creatinine clearance, albuminuria, urine N-acetyl Beta D glucosaminidase and Retinol Binding Protein, sodium clearance and sodium fractional excretion | before and after each treatment period
Other functions : blood and urine urea, total proteins, albumin, uric acid, Na+, K+, blood fasting glucose, urinary creatinine, erythrocytes, leukocytes, casts and Calculated osmolarity, free water and urinary urate | before and after each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, London, United Kingdom